CLINICAL TRIAL: NCT07250373
Title: Serratus Posterior Superior Intercostal Nerve (SPSIP) Block Versus Intercostal Nerve (ICN) Block in Patients Undergoing Uniportal Video-Assisted Thoracic Surgery (Uniportal-VATS): a Randomized Controlled Trial
Brief Title: Serratus Posterior Superior Intercostal Plane (SPSIP) Block Versus Intercostal Nerve (ICN) Block in Patients Undergoing Uniportal-VATS.
Acronym: SPUV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7594
Record Dates: First submitted 2025-06-09; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-06

CONDITIONS: Uniportal-VATS; Lung Resection Procedures; Locoregional Anesthesia; Post-operative Pain Management; Serratus Posterior Superior Intercostal Plane Block; Intercostal Nerve Block; Uniportal Video Assisted Thoracic Surgery
Keywords: SPSIP block; ICN block; Uniportal-VATS

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPSIP group (Experimental): Patients in this group will be treated with the Serratus Posterior Superior Intercostal Plane Block, administered under ultrasound guidance by the attending anesthesiologist immediately after skin closure and before extubation .
  Interventions: Other: SPSIP block
- ICN group (Active Comparator): Patients in this group will be treated with the ICN block, administered by the surgeon under direct vision at the end of surgery and immediately before skin closure.
  Interventions: Other: ICN block

INTERVENTIONS:
Other: SPSIP block — While the patient is in the lateral decubitus position, a high-frequency linear transducer is placed transversely at the level of the scapular spine, visualizing the upper medial border of the scapula, trapezius muscle, rhomboid major, serratus posterior superior muscle, and the second and third ribs. Next, the transducer is rotated to obtain an oblique view, including the upper medial border of the scapula. The needle is then advanced immediately medial to the scapula, aiming for the area between the second and third ribs to reach the fascial plane between the serratus posterior superior muscle and intercostal muscles using the in-plane technique. Once the needle contacts the rib, 30 mL of local anesthetic is administered superficially to the intercostal muscle.
  Arms: SPSIP group
Other: ICN block — The ICN block will be performed by the surgeon under direct vision at the end of surgery, immediately after skin closure, by injecting 4-5 ml of local anesthetic into the intercostal spaces from levels III-IV to VII-VIII.
  Arms: ICN group

SUMMARY:
This study aims to assess the effectiveness of the Serratus Posterior Superior Intercostal Plane (SPSIP) block compared to the Intercostal Nerve (ICN) block for postoperative pain control, reduction of opioid analgesic consumption, minimization of postoperative respiratory complications, and enhancement of patient satisfaction (measured using the QoR-15 index) in patients undergoing Uniportal Video-Assisted Thoracic Surgery (Uniportal VATS).

DETAILED DESCRIPTION:
Patients enrolled in the study will be divided into two groups: the SPSIP group and the ICN group. Patients in the SPSIP group will receive the Serratus Posterior Superior Intercostal Plane (SPSIP) block , while those in the ICN group will receive the Intercostal Nerve (ICN) block. Both blocks will be performed at the end of surgery: the SPSIP block will be administered by the attending anesthesiologist (Investigator 1) under ultrasound guidance immediately after skin closure and before extubation, while the ICN block will be performed by the surgeon under direct vision immediately before skin closure.

All patients will receive 1000 mg of paracetamol and 30 mg of ketorolac at the end of surgery, during skin closure. Upon arrival in the recovery room, each patient will be connected to a patient-controlled analgesia (PCA) pump containing an opioid-based solution. Patients reporting a Numeric Pain Rating Scale (NPRS) score greater than 4 during postoperative reassessments, despite PCA use, will be administered a rescue analgesic dose of 1000 mg of paracetamol (repeatable after 8 hours, with a maximum of 3000 mg in 24 hours).

Postoperative pain intensity will be assessed by another investigator (Investigator 2) at 0, 2, 6, 12, and 24 hours after surgery using the NPRS, both at rest and during coughing. Total opioid consumption, rescue analgesic use, incidence of postoperative complications, and length of hospital stay will also be recorded.

Twenty-four hours after surgery, Investigator 2 will administer the Quality of Recovery-15 (QoR-15) questionnaire to all patients. The responses will be used to calculate the QoR-15 index, summarizing overall patient satisfaction. Both patients and Investigator 2 will be blinded to the type of block administered, ensuring the study is conducted in a blinded manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with lung neoplasm who are candidates for pulmonary resection surgery via Uniportal-VATS
* Patients who have provided informed consent to participate in the study

Exclusion Criteria:

* Patients who refuse to participate in the study by not signing the informed consent;
* Patients with severe obesity (BMI > 35), history of OSAS with or without CPAP;
* Patients classified as ASA > 3, according to the system established by the American Society of Anesthesiologists;
* Patients unable to understand the use of the NPR Scale or the PCA device that will be used for postoperative analgesia;
* Patients with allergies to analgesic and/or anesthetic drugs;
* Patients undergoing anticoagulant therapy;
* Patients with a history of chronic pain;
* Patients with an infection at the site where SPSIPB or ICNB will be performed;
* Patients with a history of thoracic surgery and/or thoracic trauma with rib fractures on the side of surgery;
* Patients with chest wall deformities and/or neuromuscular diseases that interfere with normal ventilatory function.

Additionally, patients whose surgical procedure is intraoperatively converted to an open pulmonary resection will be excluded post hoc from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | - immediately after the end of surgery; - 2 hours after the end of surgery; - 6 hours after the end of surgery; - 12 hours after the end of surgery; - 24 hours after the end of surgery.
  The measurement of postoperative pain intensity, assessed using the Numeric Pain Rating Scale (NPRS), a numerical scale that can range from 0 to 10 (where 0 means no pain and 10 corresponds to the worst imaginable pain), in the two study groups.

SECONDARY OUTCOMES:
Total opioid drug consumption | 24 hours after the end of surgery.
  The total number of opioid doses administered via a Patient Controlled Analgesia (PCA) device in the first 24 hours after surgery
Consumption of rescue analgesics | 24 hours after the end of surgery.
  The total dose of acetaminophen administered upon the patient's request during the first 24 postoperative hours
postoperative respiratory complications | 24 hours after the end of surgery
  The number of any postoperative respiratory complications in the two study groups
postoperative quality of recovery | 24 hours after surgery
  The patient's level of satisfaction measured using the QoR-15 index, a numerical parameter calculated by administering the Quality of Recovery 15 (QoR-15) questionnaire..The QoR-15 score ranges from 0 to 150, with 0 indicating the poorest postoperative recovery quality and 150 the best
Length of Hospital Stay | from the end of surgery to the date of patient discharge, assessed up to 3 weeks
  The duration of postoperative hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Punzo, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS; Dania Nachira, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avci O, Gundogdu O, Balci F, Tekcan MN, Ozbey M. Efficacy of serratus posterior superior intercostal plane block (SPSIPB) on post-operative pain and total analgesic consumption in patients undergoing video-assisted thoracoscopic surgery (VATS): A double-blinded randomised controlled trial. Indian J Anaesth. 2023 Dec;67(12):1116-1122. doi: 10.4103/ija.ija_589_23. Epub 2023 Dec 13. PMID 38343684
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093
- [Background] Guerra-Londono CE, Privorotskiy A, Cozowicz C, Hicklen RS, Memtsoudis SG, Mariano ER, Cata JP. Assessment of Intercostal Nerve Block Analgesia for Thoracic Surgery: A Systematic Review and Meta-analysis. JAMA Netw Open. 2021 Nov 1;4(11):e2133394. doi: 10.1001/jamanetworkopen.2021.33394. PMID 34779845
- [Background] Nachira D, Meacci E, Petracca Ciavarella L, Chiappetta M, De Santis G, Ferretti GM, Mastromarino MG, Porziella V, Vita ML, Congedo MT, Cesario A, Ismail M, Gonzalez-Rivas D, Margaritora S. Uniportal video-assisted thoracic surgery Roman experience-a report of the first 16-month Roman experience. J Thorac Dis. 2018 Nov;10(Suppl 31):S3678-S3685. doi: 10.21037/jtd.2018.03.119. PMID 30505552
- [Background] Gonzalez-Rivas D, Paradela M, Fieira E, Velasco C. Single-incision video-assisted thoracoscopic lobectomy: initial results. J Thorac Cardiovasc Surg. 2012 Mar;143(3):745-7. doi: 10.1016/j.jtcvs.2011.07.049. Epub 2011 Aug 25. No abstract available. PMID 21868042